CLINICAL TRIAL: NCT02809027
Title: A Randomized Double-blind Placebo-controlled Trial on the Efficacy of Ginger in the Prevention of Abdominal Distention in Post Cesarean Section Patient
Brief Title: Efficacy of Ginger in the Prevention of Abdominal Distention in Post Cesarean Section Patient
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Vorapong Phupong, Professor Vorapong Phupong, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 114/59
Record Dates: First submitted 2016-06-16; First posted 2016-06-22 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Post Cesarean Section Patient
MeSH Terms: interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ginger (Active Comparator): Ginger capsule (500 mg), oral form, 2 capsules 3 time after meal for 3 days
  Interventions: Drug: Ginger
- Placebo (Sham Comparator): Placebo capsule, oral form, 2 capsules 3 time after meal for 3 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ginger
  Arms: Ginger
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine ginger is effective in the prevention of abdominal distention in post Cesarean section patient.

ELIGIBILITY:
Inclusion Criteria:

* Post cesarean section women

Exclusion Criteria:

* allergic to ginger
* time of cesarean section more than 1 hour
* perform another operation such as appendectomy, cystectomy
* former use carminative drugs
* already have abdominal distention

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2016-06-01; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
incidence abdominal distention as measured by diary chart (history taking and examination) | 72 hours

SECONDARY OUTCOMES:
Maternal satisfaction as measured by questionaire | 72 hours
Quality of life as measured by questionaire | 72 hours
nausea vomiting as measured by questionaire | 72 hours
first time to pass flatus/feces as measured by diary chart | 72 hours
number of carminative drug use as measured by questionaire | 72 hours
side effect as measured by questionaire | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Vorapong Phupong, M.D., Study Director — Chulalongkorn University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carroll J, Alavi K. Pathogenesis and management of postoperative ileus. Clin Colon Rectal Surg. 2009 Feb;22(1):47-50. doi: 10.1055/s-0029-1202886. PMID 20119556
- [Background] Chaiyakunapruk N, Kitikannakorn N, Nathisuwan S, Leeprakobboon K, Leelasettagool C. The efficacy of ginger for the prevention of postoperative nausea and vomiting: a meta-analysis. Am J Obstet Gynecol. 2006 Jan;194(1):95-9. doi: 10.1016/j.ajog.2005.06.046. PMID 16389016
- [Background] O'Hara M, Kiefer D, Farrell K, Kemper K. A review of 12 commonly used medicinal herbs. Arch Fam Med. 1998 Nov-Dec;7(6):523-36. doi: 10.1001/archfami.7.6.523. PMID 9821826
- [Background] Ushiroyama T, Sakuma K, Souen H, Nakai G, Morishima S, Yamashita Y, Kamegai H. Xiong-gui-tiao-xue-yin (Kyuki-chouketsu-in), a traditional herbal medicine, stimulates lactation with increase in secretion of prolactin but not oxytocin in the postpartum period. Am J Chin Med. 2007;35(2):195-202. doi: 10.1142/S0192415X07004734. PMID 17436360
- [Result] Gibstein A, Cooper JJ, Wisot AL, Rosenthal AH. Prevention of postoperative abdominal distention and discomfort with simethicone. Obstet Gynecol. 1971 Sep;38(3):386-90. No abstract available. PMID 4937581
- [Result] Hu ML, Rayner CK, Wu KL, Chuah SK, Tai WC, Chou YP, Chiu YC, Chiu KW, Hu TH. Effect of ginger on gastric motility and symptoms of functional dyspepsia. World J Gastroenterol. 2011 Jan 7;17(1):105-10. doi: 10.3748/wjg.v17.i1.105. PMID 21218090